CLINICAL TRIAL: NCT04427241
Title: Efficacy and Safety of Cerebrolysin on Prolonged Disorders of Consciousness in Patients With Hemorrhagic Stroke: A Pilot Study
Brief Title: Efficacy and Safety of Cerebrolysin on Prolonged Disorders of Consciousness
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Konkuk University Medical Center (Other)
Collaborators: Ever Neuro Pharma GmbH (Industry)
Responsible Party: Principal Investigator, Jongmin Lee, MD, PhD, Professor, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: kuhrm2020no1
Record Dates: First submitted 2020-06-03; First posted 2020-06-11 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Disorder of Consciousness; Hemorrhagic Stroke
MeSH Terms: conditions — Consciousness Disorders; Hemorrhagic Stroke | interventions — cerebrolysin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cerebrolysin (Experimental): 30 ml cerebrolysin + 70 ml normal saline, days 4-17, once/day, intravenously
  Interventions: Drug: Cerebrolysin
- Control (Placebo Comparator): 100 ml normal saline, days 4-17, once/day, IV
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Cerebrolysin — 30 ml cerebrolysin + 70 ml normal saline, days 4-17, once/day, intravenously
  Arms: Cerebrolysin
Drug: Control — 100 ml normal saline, days 4-17, once/day, IV
  Arms: Control

SUMMARY:
Object: To determine the effect of cerebrolysin on prolonged disorders of consciousness caused by hemorrhagic stroke.

Participants: patients with prolonged disorders of consciousness due to severe traumatic brain injury

Intervention: 30 ml cerebrolysin + 70 ml normal saline, days 4-17, once/day, intravenously or 100 ml normal saline, days 4-17, once/day, IV

Comparison: cerebrolysin group versus control group

Outcome: Coma Recovery Scale-revised, FDG-PET signal

ELIGIBILITY:
Inclusion Criteria

1. Patients with hemorrhagic stroke confirmed by CT or MRI
2. Patients who have been in disorders of consciousness for more than 4 weeks after the onset of hemorrhagic stroke
3. Patients in a vegetative state or minimally conscious state (Coma Recovery Scale -revised: CRS-R assessment)
4. Age: 19 to 80 years of age
5. Patients who have voluntarily given written informed consent to participate in the study by themselves or their legal representative.

Exclusion Criteria

1. Patients with confirmed epileptiform discharges on EEG
2. Patients with brain parenchymal defects
3. Patients with advanced liver, kidney, cardiac, or pulmonary disease.
4. Chronic treatment with medications that may affect consciousness, such as antidepressants, antipsychotic drugs, nootropic drugs, and vasodilators.
5. History of serious illness within the last two years (cancer, hematologic, renal, hepatic, or coronary artery disease, psychiatric illness, diabetes, myocardial infarction, epilepsy), no evidence of secondary damage to major organs, and well-controlled diabetes or hypertension.
6. Alcohol or drug abuse or dependence within the last 2 years (DSM-V criteria).
7. Significant systemic disease or unstable medical condition that may compromise compliance with the study protocol.
8. Administration of a contraindicated drug is essential for medical purposes.
9. Contraindications to the study drug (cerebrolysin).
10. Participation in another therapeutic study

Ages: 19 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Coma Recovery Scale - revised | 2 days after randomization
  Assessing the degree of disorders of consciousness
Coma Recovery Scale - revised | 17 days after randomization
  Assessing the degree of disorders of consciousness
Positron Emitting Tomography | 2 days after randomization
  Assessing the degree of brain neural network activity
Positron Emitting Tomography | 17 days after randomization
  Assessing the degree of brain neural network activity

CONTACTS AND LOCATIONS:
Locations (1):
- Konkuk University Medical Center Research Coordinating Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee S, Lee HH, Lee Y, Lee J. Additive effect of cerebrolysin and amantadine on disorders of consciousness secondary to acquired brain injury: A retrospective case-control study. J Rehabil Med. 2020 Feb 27;52(2):jrm00025. doi: 10.2340/16501977-2654. PMID 32057086
- [Background] Giacino JT, Whyte J, Bagiella E, Kalmar K, Childs N, Khademi A, Eifert B, Long D, Katz DI, Cho S, Yablon SA, Luther M, Hammond FM, Nordenbo A, Novak P, Mercer W, Maurer-Karattup P, Sherer M. Placebo-controlled trial of amantadine for severe traumatic brain injury. N Engl J Med. 2012 Mar 1;366(9):819-26. doi: 10.1056/NEJMoa1102609. PMID 22375973